CLINICAL TRIAL: NCT04364789
Title: A Phase I, First-In-Human, Randomized, Double-blind, Placebo-controlled, Single-Ascending-Dose Study of TT-00920 in Healthy Subjects
Brief Title: Phase I, First-In-Human Study of TT-00920 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TransThera Sciences (Nanjing), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TT00920US01
Record Dates: First submitted 2020-04-21; First posted 2020-04-28 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Paticipant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Pilot dose Cohort (Active Comparator): A pilot dose of 20 mg will be evaluated in 2 subjects (all receiving TT-00920) for safety, tolerability, and PK profile before the initiation of dose escalation.
  Interventions: Drug: TT-00920
- SAD Dose 1 (Active Comparator)
  Interventions: Drug: TT-00920
- SAD Dose 2 (Active Comparator)
  Interventions: Drug: TT-00920
- SAD Dose 3 (Active Comparator)
  Interventions: Drug: TT-00920
- SAD Dose 4 (Active Comparator)
  Interventions: Drug: TT-00920
- Food Effect Cohort (Active Comparator)
  Interventions: Drug: TT-00920
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: TT-00920 — Tablets
  Arms: Food Effect Cohort; Pilot dose Cohort; SAD Dose 1; SAD Dose 2; SAD Dose 3; SAD Dose 4
Drug: Placebos — Tablets
  Arms: Placebo

SUMMARY:
This is a first-in-human, randomized, double-blind, placebo-controlled study. The primary objectives of the study were to investigate the safety and tolerability and determine the PK profiles of single ascending doses (SAD) of TT-00920 administered to healthy subjects. The secondary objectives of the study were to assess the effect of food on the PK of TT-00920 following an oral dose.

DETAILED DESCRIPTION:
There will be 4 single-ascending-dose cohorts and 1 cohort for food effect assessment to assess the safety, tolerability, and PK profile. A pilot dose of 20 mg will be evaluated in 2 subjects (all receiving TT-00920) for safety, tolerability, and PK profile before the initiation of dose escalation.

In single-ascending-dose cohorts, 8 subjects per cohort will be enrolled and randomized to assess the safety, tolerability, and PK profile. In food effect cohort, there will be 8 subjects (all receiving TT-00920). Subjects in food effect cohort will receive 2 single dose periods (Fasted/ Fed) in an open-label, crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Age ≥ 18 years and ≤ 55 years, male or female of non-childbearing potential (confirmed with follicle stimulating hormone [FSH] test. A bilateral tubal ligation is acceptable as long as there is no fertility potential).
* Body mass index (BMI) between 18 and 30 kg/m2, inclusive, and weighs at least 50 kg.
* No clinically significant findings in medical examination

Exclusion Criteria:

* Any history of clinically serious disease.
* Hypersensitivity or allergy to any of the study drugs or drugs of similar chemical classes.
* Impaired cardiac function including clinically significant arrhythmias or clinically significant abnormality in clinical test
* Subject with a history of severe visual diseases; or visual changes including flushing lights, blurry vision, color changes, or other visual changes; or abnormal finding with visual tests [color discrimination (Ishihara test) and visual acuity (Snellen chart).
* Subject is unable to complete this study for other reasons or the Investigator believes that he or she should be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Numbers of Treatment Emergent Adverse Events(TEAE) | 10 days
  Safety and tolerability of TT-00920
Number of participants with Abnormal Laboratory Values | 10 days
  Safety and tolerability of TT-00920
Area under the plasma drug concentration versus time curve | 10 days
  PK parameters of TT-00920
Maximum Observed Plasma Concentration (Cmax) | 10 days
  PK parameters of TT-00920
Time of First Occurrence of Cmax （tmax) Time of first Occurance of Cmax（tmax) | 10 days
  PK parameters of TT-00920
Terminal half-life (t1/2) | 10 days
  PK parameters of TT-00920
Elimination rate (λz) | 10 days
  PK parameters of TT-00920
Volume of distribution (Vz/F) | 10 days
  PK parameters of TT-00920
Clearance (CL/F) | 10 days
  PK parameters of TT-00920

SECONDARY OUTCOMES:
Area under the plasma drug concentration versus time curve | 10 days
  the effect of food on the PK of TT-00920 following an oral dose
Maximum Observed Plasma Concentration (Cmax) | 10 days
  the effect of food on the PK of TT-00920 following an oral dose
Time of first Occurance of Cmax（tmax) | 10 days
  the effect of food on the PK of TT-00920 following an oral dose
Terminal half-life (t1/2) | 10 days
  the effect of food on the PK of TT-00920 following an oral dose
Elimination rate (λz) | 10 days
  the effect of food on the PK of TT-00920 following an oral dose
Volume of distribution (Vz/F) | 10 days
  the effect of food on the PK of TT-00920 following an oral dose
Clearance (CL/F) | 10 days
  the effect of food on the PK of TT-00920 following an oral dose

OTHER OUTCOMES:
Metabolite characterization in plasma and estimation of observed drug-related material in plasma to determine the presence of any metabolite >10% | 10 days
  Exploratory outcome measures
Cyclic guanosine monophosphate (cGMP) levels in plasma and urine | 10days
  Exploratory outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: Gevorkyan Hakop, MD, Principal Investigator — Early Phase Clinical Unit Glendale Adventist Medical Center
Locations (1):
- Early Phase Clinical Unit Glendale Adventist Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No